CLINICAL TRIAL: NCT03393039
Title: Neural Effects of Negative Affect on Food Choices and Reward In Individuals With Binge Eating Episodes
Brief Title: Effects of Negative Affect in Individuals With Binge Eating Episodes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Sanford Research (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-2658
Record Dates: First submitted 2017-12-28; First posted 2018-01-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder; Obesity; Eating Disorder
Keywords: fMRI; Reward; Food Choices; Negative Affect
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral (Experimental): Negative Affect Task
  Interventions: Behavioral: Negative Affect Task

INTERVENTIONS:
Behavioral: Negative Affect Task — fMRI stress task
  Other Names: Functional Magnetic Resonance Brain Imaging Stress Task

SUMMARY:
Binge-eating is characterized by recurrent episodes of eating large amounts of - typically high calorie - foods, eating much more rapidly than normal and until feeling uncomfortably full, as well as feeling disgusted with oneself, depressed, or guilty after those episodes. Two eating disorders are characterized by binge-eating as central diagnostic criteria, binge-eating disorder (BED) and bulimia nervosa (BN). Binge-eating episodes in BN, but not BED, are typically followed by compensatory mechanisms such as self-induced vomiting, and BED is typically associated with obesity, while BN is not. Behavior studies such as ecological momentary assessment (EMA) research of affect in an individual's naturalistic environment have shown that negative affect and negative urgency (the tendency to act rashly when distressed) often precede binge-eating.

The Investigators want to answer the following questions: Can negative affect in BN and BED be linked to 1) altered dopamine related brain reinforcement learning, 2) to food value computation and cognitive control circuit function, and 3) can dopamine related brain activation predict eating and negative affect, indicating a brain based neurobiological vulnerability. Answering those questions will help to define binge-eating based on regulation of brain reward, cognition, and emotion circuit function and point toward potential psychopharmacological interventions to normalize brain function and behavior.

DETAILED DESCRIPTION:
Specific Aim 1: To test on two study days, one neutral affect and one negative affect day (affect induction) whether negative affect alters brain reinforcement learning in a dopamine system anchored taste reward learning paradigm (a task for prediction error and reward value computation) during functional magnetic resonance brain imaging (fMRI). Hypothesis 1: In response to negative and compared to neutral affect induction, binge eating disorder (BED) and bulimia nervosa (BN) will show increased positive prediction error and taste valuation regression with striatum and insula activation compared to obese (OB) and healthy control (HC) groups. This will be an indication that negative affect excessively activates dopamine related reward circuit response in BED and BN. Specific Aim 2: To study during a food choice paradigm the effects of negative affect on brain circuitry for cognitive control and food valuation. Specific Aim 2a: To study brain circuitry for food valuation in response to neutral or negative affect. Hypothesis 2a: In response to negative and compared to neutral affect induction, BED and BN groups will show greater striatal activation when rating food for taste, compared to OB and HC. This will indicate that BED and BN are associated with increased affect-regulated motivation to approach high calorie foods after negative affect induction and compared to OB and HC. Specific Aim 2b: To study brain control circuitry during food choice in response to neutral or negative affect. Hypothesis 2b: In response to negative and compared to neutral affect induction, BED and BN groups will show increased insula and striatal, but lower dorsolateral prefrontal cortex (DLPFC) activation compared to OB and HC groups. This will indicate that negative affect activates automatic food reward circuit response, but reduces cognitive control circuitry during food choice in BED and BN. Specific Aim 3: To test whether brain activation predicts food intake or negative affect. Specific Aim 3a: To test whether brain activation can predict food intake during a post-fMRI scan test meal. Hypothesis 3a: On negative- versus neutral-affect days, BN and BED will select more food in a post-fMRI scan test meal; lower DLPFC and higher striatal activation during food choice, and higher (prediction error) taste reward activation in insula and ventral striatum will predict greater food intake. Specific Aim 3b: To test whether brain activation during reward learning or food choice predicts negative affect measured by EMA on the study day, as well as measured between study days in the individual's naturalistic environment. Hypothesis 3b: Insula, ventral striatum and DLPFC activation (taste prediction error task, food choice task) during the negative affect condition will predict the intensity of negative affect immediately after fMRI, as well as intensity of negative affect episodes during the days between brain scans in the individual's naturalistic environment, suggesting a neurobiological affective vulnerability.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* Age 18-55 years old
* Healthy body weight between 90 and 110 % average body weight since puberty.
* Regular monthly menstrual cycle (if applicable)
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200

Obese

* Age 18-55 years old
* Current body mass index (BMI) > 30 kg/m2.
* Stable food intake regimen in previous 4 weeks.
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* Obese for at least one year

Binge Eating Disorder

* Age 18-55 years old
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* DSM 5 diagnosis of Binge Eating Disorder A. Recurrent episodes of binge eating B. Binge eating episodes are associated with three (or more) of the following

  1. Eating much more rapidly than normal.
  2. Eating until feeling uncomfortably full.
  3. Eating large amounts of food when not feeling physically hungry.
  4. Eating alone because of embarrassment.
  5. Feeling disgusted with oneself, depressed, or very guilty after overeating. C. Marked distress regarding binge eating is present. D. At least once a week for 3 months. E. The binge eating is not associated with the recurrent use of inappropriate compensatory behavior.

Bulimia Nervosa

* Age 18-55 years old
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* DSM 5 diagnosis of Bulimia Nervosa A. Recurrent episodes of binge eating Eating, in a discrete period of time, an amount of food that is definitely larger than most people would eat during a similar period of time and under similar circumstances.

A sense of lack of control over eating during the episode. B. Recurrent inappropriate compensatory behavior in order to prevent weight gain, such as self-induced vomiting; misuse of laxatives, diuretics, or other medications; fasting; or excessive exercise.

C. At least once a week for 3 months. D. Self-evaluation is unduly influenced by body shape and weight.

Exclusion Criteria:

Healthy Controls

* Current pregnancy or breast feeding within last 3 months
* First degree relative with current or past eating disorder
* Current Medications other than BCP or IUD
* Past or present Axis I psychiatric disorder including substance or alcohol use disorder as determined through SCID-5 clinical interview
* First degree relative with an eating disorder
* Major Medical illness
* Recent history of suspected substance abuse or a lifetime history of psychostimulant abuse and/or dependence
* Metal implants or braces

Obese

* Current pregnancy or breast feeding within last 3 months
* First degree relative with current or past eating disorder
* Current or previous eating disorder diagnosis
* Current Medications other than BCP or IUD
* Past or present Axis I psychiatric disorder including substance or alcohol use disorder as determined through SCID-5 clinical interview
* Major Medical illness
* Recent history of suspected substance abuse or a lifetime history of psychostimulant abuse and/or dependence
* Metal implants or braces

Binge Eating Disorder

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar disorder or psychosis
* Use of a psychostimulant within the prior 6 months
* Recent history of substance abuse or dependence (except for alcohol and cannabis use)
* Major Medical illness
* Metal implants or braces

Bulimia Nervosa

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar disorder or psychosis
* Use of a psychostimulant within the prior 6 months
* Recent history of substance abuse or dependence (except for alcohol and cannabis use)
* Major Medical illness
* Metal implants or braces

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 410 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Taste Reward Brain Response to Negative Affect fMRI Task | 5 years
  to study brain activation in a taste reward task in response to negative affect
Food Choice Brain Response to Negative Affect fMRI Task | 5 years
  to study brain activation in a food choice task in response to negative affect
Brain Activation and Food Intake/negative Affect Relationships | 5 years
  To test whether brain activation predicts food intake or negative affect

CONTACTS AND LOCATIONS:
Overall Officials: Guido KW Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California at San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Engel SG, Kahler KA, Lystad CM, Crosby RD, Simonich HK, Wonderlich SA, Peterson CB, Mitchell JE. Eating behavior in obese BED, obese non-BED, and non-obese control participants: a naturalistic study. Behav Res Ther. 2009 Oct;47(10):897-900. doi: 10.1016/j.brat.2009.06.018. Epub 2009 Jul 7. PMID 19631931
- [Background] Berg KC, Crosby RD, Cao L, Crow SJ, Engel SG, Wonderlich SA, Peterson CB. Negative affect prior to and following overeating-only, loss of control eating-only, and binge eating episodes in obese adults. Int J Eat Disord. 2015 Sep;48(6):641-53. doi: 10.1002/eat.22401. Epub 2015 Mar 23. PMID 25808854
- [Background] Pearson CM, Wonderlich SA, Smith GT. A risk and maintenance model for bulimia nervosa: From impulsive action to compulsive behavior. Psychol Rev. 2015 Jul;122(3):516-35. doi: 10.1037/a0039268. Epub 2015 May 11. PMID 25961467
- [Background] Racine SE, Burt SA, Keel PK, Sisk CL, Neale MC, Boker S, Klump KL. Examining associations between negative urgency and key components of objective binge episodes. Int J Eat Disord. 2015 Jul;48(5):527-31. doi: 10.1002/eat.22412. Epub 2015 Apr 10. PMID 25865091
- [Background] Engel SG, Crosby RD, Thomas G, Bond D, Lavender JM, Mason T, Steffen KJ, Green DD, Wonderlich SA. Ecological Momentary Assessment in Eating Disorder and Obesity Research: a Review of the Recent Literature. Curr Psychiatry Rep. 2016 Apr;18(4):37. doi: 10.1007/s11920-016-0672-7. PMID 26893235